CLINICAL TRIAL: NCT01117545
Title: Psychological Symptom Change in Veterans After Six Sessions of EFT (Emotional Freedom Techniques): A Randomized Controlled Trial
Brief Title: Psychological Symptom Change in Veterans After Six Sessions of EFT (Emotional Freedom Techniques)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SMI-PTSD-5410
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: veterans,; PTSD,; EFT (Emotional Freedom Techniques),; depression,; anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFT (Experimental): Six sessions of EFT (Emotional Freedom Techniques)
  Interventions: Behavioral: EFT (Emotional Freedom Techniques)
- Wait List (No Intervention): One month wait period

INTERVENTIONS:
Behavioral: EFT (Emotional Freedom Techniques) — Six sessions of EFT
  Arms: EFT

SUMMARY:
EFT (Emotional Freedom Techniques) has been shown to significantly reduce post-traumatic stress disorder (PTSD) and other psychological symptoms such as anxiety and depression in a variety of clinical trials. This study examines the effect of a six session EFT protocol on the symptoms of veterans with clinical scores on the PTSD Checklist-Military (PCL-M). Subjects in the experimental group receive EFT coaching supplemental to, and supportive of, the "usual care" treatment provided by their primary care provider. Subjects in the wait list control group receive usual care for a month, with pre and posttests, after which they also receive the EFT coaching protocol. Subjects are followed at three month intervals to determine if gains are maintained, and whether the symptom reductions are similar to those observed in other trials of EFT.

ELIGIBILITY:
Inclusion Criteria:

* Military Service
* The ability to follow instructions, complete written forms, and provide informed consent.
* Remaining under the care of a primary care provider such as a VA hospital throughout the entire period of the study
* Between 18 and 90 years old

Exclusion Criteria:

* Participants with a score of more than 3 on questions 34 and 35 of the Symptom Assessment-45 Questionnaire (SA-45) will receive phone/skype sessions, not office visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
PTSD Scores on the PCL-M Assessment | One Month Before, At Start, After 3 and 6 Sessions, After 3 and 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- [Result] Church D, Hawk C, Brooks AJ, Toukolehto O, Wren M, Dinter I, Stein P. Psychological trauma symptom improvement in veterans using emotional freedom techniques: a randomized controlled trial. J Nerv Ment Dis. 2013 Feb;201(2):153-60. doi: 10.1097/NMD.0b013e31827f6351. PMID 23364126
- See also: Veterans Stress Project. This site is a primary web site recruiting subjects. — http://www.StressProject.org